CLINICAL TRIAL: NCT05397210
Title: Post-market Clinical Follow-up (PMCF) Study of the Infinity-Lock™ Button System for Acromioclavicular Joint Stabilisation
Brief Title: Post-market Clinical Follow-up (PMCF) Study of the Infinity-Lock Button System for Acromioclavicular Joint Stabilisation
Status: Recruiting | Type: Observational
Sponsor: Xiros Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CRE 019
Record Dates: First submitted 2022-05-24; First posted 2022-05-31 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Acromioclavicular; Dislocation
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Infinity-Lock™ Button System: Participants diagnosed with acute or chronic Grade Ill-VI ACJ dislocation who require treatment with an Infinity-Lock Button System who meet the inclusion criteria and none of the exclusion criteria.
  Interventions: Device: Infinity-Lock Button System

INTERVENTIONS:
Device: Infinity-Lock Button System — Infinity-Lock Button System

SUMMARY:
This is a Post-market Clinical Follow-up Study. It will verify the long-term safety and performance of the Infinity-Lock Button System (ILBS) when used for acute and chronic dislocations of the Acromioclavicular Joint and used as described by the manufacturer's instructions.

DETAILED DESCRIPTION:
This is a Post-market Clinical Follow-up Study. It will verify the long-term safety and performance of the Infinity-Lock Button System (ILBS) when used for acute and chronic dislocations of the Acromioclavicular Joint and used as described by the manufacturer's instructions.

The medical device (ILBS) in this study is already on the market and is manufactured by Xiros Ltd.

The ILBS comprises of a polyester flexible tubular tape and a titanium button. The tape is used to secure the joint and the button is used to secure the tape into position.

This study will collect data on patients who meet the entry criteria and receive the device; it will recruit patients from several clinical sites.

All patients in the study will receive the ILBS, as it is a single armed study. The total length of the study is expected to be 4.5 years; this includes a recruitment period of approximately 18 months and a 3-year follow-up.

A total of 58 subjects will be enrolled into the study. Follow up is at 3 months, 6 months, 1,2 and 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 16 years old or above.

  * Patient is diagnosed with acute or chronic Grade Ill-VI ACJ dislocation.
  * Patient is willing to participate in the study and have been informed of the nature of the study, agree to its follow-up and have provided written informed consent as approved by the Research Ethics Committee (REC).

Exclusion criteria.

* Known hypersensitivity to implant materials. If the patient is suspected of having any foreign body sensitivity, appropriate tests should be made prior to implantation.
* Infections or any other structural or pathological condition of the bone or soft tissue (such as hyperlaxity) that would be expected to impair healing or secure fixation.
* Patients unable or unwilling to restrict activities to prescribed levels or follow a rehabilitation programme during the healing period.
* Skeletally immature patients are not suited as the Infinity-Lock™ Button System will not elongate with growth. The use of this medical device and placement of hardware or implants must not bridge, disturb or disrupt the growth plate.
* Any other conditions or factors which in the opinion of the Investigator may interfere with study conduct.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Grade III-VI ACJ Dislocations.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Constant Murley Score (CMS) | 1 year
  The primary performance endpoint is the change in the CMS from baseline to 1 year after surgery. Minimum score is 0 maximum is 100 with the better functioning shoulders having a greater number of points.
Device Related or Procedure Related Adverse events | 1 year
  device-related and/or procedure-related adverse events up to 1 year after surgery.

SECONDARY OUTCOMES:
Constant Murley Score (CMS) | 3 years
  Change from baseline CMS and subscale scores (pain, activities of daily living, strength and ROM) at each timepoint up to 3 years after surgery. Minimum score is 0 maximum is 100 with the better functioning shoulders having a greater number of points.
American Shoulder and Elbow Surgeons Score (ASES) | 3 years
  Change from baseline American Shoulder and Elbow Surgeons (ASES) Score at each timepoint up to 3 years after surgery. Total score 0-100 ASES points, 0 = worse pain and functional loss/disability.
RAND Short Form 36 (SF-36) V1 | 3 years
  Change from baseline RAND Short Form 36 (SF-36) V1 Quality of Life Health Survey at each timepoint up to 3 years after surgery.The RAND SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Nottingham Clavicle Score (NCS) | 3 years
  Change from baseline Nottingham Clavicle Score (NCS) at each timepoint up to 3 years after surgery. Maximum score of 100 (fewest difficulties) and a minimum score of 20 (most difficulties)
Ability to perform normal daily work and normal recreational activities | 3 years
  This is a subscale of the CMS and is a measurement of how much of the normal daily work or recreational activity the patient is able to perform. The scale is a line which will be marked by the subject, it will be reported as 0-100% with 100% meaning they are able to perform 100% of their normal daily work or recreational activity
coracoclavicular distance | 1 year
  Change from baseline CC distance using the anteroposterior (AP) X-ray (Zanca view) at each timepoint up to 1 year after surgery.
Device-related and/or procedure-related adverse events | 3 years
  Device-related and/or procedure-related adverse events up to 3 years after surgery.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - East Kent Hospitals University NHS Foundation Trust,, Canterbury
  - Barts Health NHS Trust, London
  - Nottingham University Hospitals, Nottingham
  - Royal Berkshire NHS Foundation Trust, Reading

IPD SHARING:
Plan to Share IPD: No
No plan to share IDP